CLINICAL TRIAL: NCT00396708
Title: Wearable Robotic Functional Assistance for Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Myomo (Industry)
Responsible Party: Kailas Narendran, Myomo,Inc
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2006-11-03; First posted 2006-11-07 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: CVA (Cerebrovascular Accident)
Keywords: Robotics; Rehabilitation; Arm; Stroke; Weakness; Outpatient; Chronic
MeSH Terms: conditions — Stroke; Asthenia; Bronchiolitis Obliterans Syndrome

INTERVENTIONS:
Device: myomo e100 neurorobotic elbow brace

SUMMARY:
This study aims to evaluate the effectiveness of using the myomo e100 wearable robotic rehabilitation system for increasing functional independence and long term rehabilitation of chronic stroke victims with a hemiparetic upper extremity.

DETAILED DESCRIPTION:
This is a case controlled study for evaluation of the effectiveness of using the myomo e100 wearable robotic rehabilitation for upper arm therapy following stroke.

The intervention for the study will be for the control group- 6-8 weeks of therapeutic exercise and functional training for a total of 18 hours of intervention, or the case group- 6-8 weeks of therapeutic exercise and functional training with the use of the AJB for a total of 18 hours of intervention. Each session will be one hour in length. The length of the study and length of each session is per standard rehabilitation protocol that has been well documented in previous studies as well as the pilot study regarding the AJB. A pre and post test with a 3 month follow up of all measures will be included in the study.

Study procedures will focus on performing functional tasks using the e100.

ELIGIBILITY:
Inclusion Criteria:

* Medically Stable
* Cognitive Awareness
* Weakness in upper arm
* Over 1 year post CVA
* not engaged in any other upper arm therapies

Exclusion Criteria:

* Rashes, open wounds or skin sensitivity on arm
* Very high elbow tone (arm rigid in flexion or extension)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-08; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Motor Activity Log
Fugl-Meyer Upper Arm Function
Wolf Motor Function
SF-36 QOL Survey
Range of Motion
Muscle Strength Test

CONTACTS AND LOCATIONS:
Overall Officials: Kailas N Narendran, BS, MEng, Principal Investigator — Inventor
Locations (1):
- myomo Inc., Boston, Massachusetts, United States

REFERENCES:
- See also: Myomo Inc. Homepage — http://www.myomo.com/